CLINICAL TRIAL: NCT00577655
Title: Phase 3 Study to Evaluate the Chronic-dose Safety and Efficacy of Albuterol-HFA-MDI Relative to Placebo in Pediatric Asthmatics
Brief Title: Albuterol HFA MDI in Pediatric Participants With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IXR-302-25-105
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: Pediatric, asthma, albuterol-HFA and Placebo
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albuterol (Experimental): Albuterol-HFA-MDI 180 mcg, four times a day (total daily albuterol dose of 720 mcg) for 21 days. HFA-MDI refers to a metered-dose inhaler (MDI) utilizing a hydrofluoroalkane (HFA) propellant.
  Interventions: Drug: Albuterol; Drug: Proventil® HFA
- Placebo (Placebo Comparator): A placebo of a metered-dose inhaler (MDI) utilizing a hydrofluoroalkane (HFA) propellant. (Hereafter noted as "Placebo-HFA-MDI.")
  Interventions: Drug: Placebo; Drug: Proventil® HFA

INTERVENTIONS:
Drug: Albuterol — Albuterol HFA MDI 180 mcg four times a day (q.i.d) for a total daily albuterol dose of 720 mcg for 21 days.
  Other Names: ProAir® HFA; Albuterol Sulfate
  Arms: Albuterol
Drug: Placebo — Placebo HFA MDI four times a day (q.i.d) for 21 days.
  Arms: Placebo
Drug: Proventil® HFA — Proventil® HFA (albuterol sulfate) Inhalation Aerosol (Key Pharmaceuticals) was used as rescue medication in this study. The rescue medication was over-labeled with instructions for emergency use in which subjects were instructed to self-administer up to two puffs every 20 minutes to a maximum of six puffs for any given episode while attempting to seek medical assistance.
  Other Names: albuterol sulfate

SUMMARY:
The primary objective of this study is to evaluate the chronic-dose and efficacy of Albuterol-HFA-MDI relative to placebo in pediatric asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female child aged 4-11 years, inclusive Asthma of a minimum of six months duration that has been stable for at least four weeks prior to screening.

Exclusion Criteria:

* Hospitalization for acute asthma exacerbation greater than two years in 12 months prior to screening and/or received ER treatment or hospitalization for asthma exacerbation.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Study Physician MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (13):
- United States (13):
  - Pediatric Care Medical Group, Inc., Huntington Beach, California
  - California Allergy & Asthma Medical Group, Palmdale, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Integrated Research Group, Inc, Riverside, California
  - Center for Clinical Trials of Sacramento, Sacramento, California
  - Carlos Piniella, MD, Miami, Florida
  - Sneeze, Wheeze & Itch Associates, Inc., Normal, Illinois
  - Asthma & Allergy Associates, PC, Elmira, New York
  - ENT & Allergy Associates, Newburgh, New York
  - St. Elizabeth's Children Health Center, Utica, New York
  - Regional Allergy & Asthma Consultants, Asheville, North Carolina
  - Clinical Research Institute of Southern Oregan, PC, Medford, Oregon
  - Virginia Adult & Pediatric Allergy & Asthma, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 208 individual subjects were screened; ten subjects failed the initial screening but were later re-screened and successfully enrolled.
Groups:
- Albuterol: Albuterol-HFA-MDI 180 mcg, four times a day (total daily albuterol dose of 720 mcg) for 21 days.
- Placebo: Placebo HFA-MDI four times a day for 21 days.
Period: Overall Study
Arm/Group | Albuterol | Placebo
Started | 52 (This number represents the number of participants randomized.) | 51 (This number represents the number of participants randomized.)
Completed | 51 | 47
Not Completed | 1 | 4
Not completed — Patient Request | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Albuterol | Placebo | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.3 (1.82) | 8.2 (2.09) | 8.2 (1.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 33 | 31 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  White | 30 | 39 | 69
  Black | 14 | 7 | 21
  Asian | 5 | 3 | 8
  North American Indian or Alaska native | 1 | 1 | 2
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 52 | 51 | 103
Forced Expiratory Volume in One Second (FEV1) on Day 1 [Mean (Standard Deviation); unit: liters] — Baseline measurement is the average of two Day 1 pre-dose FEV1 values. n=51, 51, 103
  liters | 1.52 (0.38) | 1.49 (0.46) | 1.50 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Change From Baseline in Forced Expiratory Volume in One Second (FEV1) Observed up to Two Hours Post Dose (FEV1max%0-2) on Day 22
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters. A standardized spirometer was used with the subject in the sitting or standing position (orientation had to be consistent for each subject during study visits) and wearing a nose clip. Whenever possible, evaluations were performed by the same respiratory therapist on the same calibrated spirometer at approximately the same time (±2 hrs).
  The maximum percent change from baseline in FEV1 observed up to 2 hours following completion of dosing using Day 22 baseline. The baseline FEV1 was defined as the average of the two test-day pre-dose baseline FEV1 values.
  The reason for the two primary endpoints was that FEV1 is difficult to obtain in children below 7 years of age.
Time Frame: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5, 45±5, 60±10, 120 ±10 post dosing on Day 22 or last observation
Population: Intent-To-Treat (ITT) population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: percentage change from baseline
Groups:
- Placebo: Placebo-HFA-MDI four times a day for 21 days.
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
percentage change from baseline | 12.849 (1.005) | 9.353 (1.017)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Efficacy was declared if the test for either primary efficacy endpoint was significant at the 0.025 level; Test type: Superiority or Other; p = 0.0138, ANCOVA — In order to control the overall alpha level at the 0.05 value, each of the primary endpoints were tested separately at the 0.025 level of significance; Baseline as covariate and fixed effects of treatment and pooled investigator site; Mean Difference (Final Values) = 3.496, 95% CI 2-sided [0.729 to 6.262] — Active - Placebo

2. Primary Outcome: Maximum Percent Change From Baseline in Peak Expiratory Flow (PEF) Observed up to Two Hours Post Dose (PEFmax%0-2) on Day 22
Description: The PEF test is conducted by having a person blow as hard as they can into a mouthpiece attached to a sensor that measures the rate of air blown. A standardized spirometer was used with the subject in the sitting or standing position (orientation had to be consistent for each subject during study visits) and wearing a nose clip. Whenever possible, evaluations were performed by the same respiratory therapist on the same calibrated spirometer at approximately the same time (±2 hrs).
  The maximum percent change from baseline in the PEF observed up to 2 hours following completion of dosing using Day 22 baseline. The baseline PEF was defined as the average of the test-day pre-dose baseline PEF values.
  The reason for the two primary endpoints was that FEV1 is difficult to obtain in children below 7 years of age.
Time Frame: 30±5 and 5±2 minutes prior to dosing, and at 7.5±2, 20±5, 35±5, 50±5, 65±10, 125±10 post dosing on Day 22 or last observation
Population: Intent-To-Treat (ITT) population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
percentage change from baseline | 17.558 (1.878) | 12.127 (1.907)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Efficacy was declared if the test for either primary efficacy endpoint was significant at the 0.025 level; Test type: Superiority or Other; p = 0.0403, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Baseline as covariate and fixed effects of treatment and pooled investigator site; Mean Difference (Final Values) = 5.431, 95% CI 2-sided [0.244 to 10.618] — Active - Placebo

3. Secondary Outcome: Maximum Percent Change From Baseline in Forced Expiratory Volume in One Second (FEV1) up to Two Hours Post-Dose (FEV1max%0-2, %) on Study Days 1 and 22 Using Observed Cases
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters. A standardized spirometer was used with the subject in the sitting or standing position (orientation had to be consistent for each subject during study visits) and wearing a nose clip. Whenever possible, evaluations were performed by the same respiratory therapist on the same calibrated spirometer at approximately the same time (±2 hrs).
  The maximum percent change from baseline in FEV1 observed up to 2 hours following completion of dosing using test day baseline. The baseline FEV1 was defined as the average of the two test-day pre-dose baseline FEV1 values.
Time Frame: Days 1 and 22: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5, 45±5, 60±10, 120 ±10 post dosing
Population: Observed cases (i.e. available data only)
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 51 | 51
percentage change from baseline
  Day 1 (n=51, 51) | 12.621 (1.072) | 8.085 (1.075)
  Day 22 (n=51, 47) | 12.601 (1.072) | 9.534 (1.119)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1 A repeated measures mixed model, with terms for treatment, pooled center, study day, treatment by study day interaction, and baseline as a covariate, and subject as a random term, was used to make comparisons between placebo and active with respect to FEV1max%0-2 at Days 1 and 22, with observed case data; Test type: Superiority or Other; p = 0.0031, Mixed Models Analysis — significance level of 0.05; Mean Difference (Final Values) = 4.536, 95% CI 2-sided [1.567 to 7.505] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22 A repeated measures mixed model, with terms for treatment, pooled center, study day, treatment by study day interaction, and baseline as a covariate, and subject as a random term, was used to make comparisons between placebo and active with respect to FEV1max%0-2 at Days 1 and 22, with observed case data; Test type: Superiority or Other; p = 0.0470, Mixed Models Analysis — significance level of 0.05; Mean Difference (Final Values) = 3.067, 95% CI 2-sided [0.041 to 6.094] — Active - Placebo

4. Secondary Outcome: Maximum Percent Change From Baseline in Peak Expiratory Flow (PEF) up to Two Hours Post-Dose (PEFmax%0-2) on Study Days 1 and 22 Using Observed Cases
Description: The PEF test is conducted by having a person blow as hard as they can into a mouthpiece attached to a sensor that measures the rate of air blown. A standardized spirometer was used with the subject in the sitting or standing position (orientation had to be consistent for each subject during study visits) and wearing a nose clip. Whenever possible, evaluations were performed by the same respiratory therapist on the same calibrated spirometer at approximately the same time (±2 hrs).
  The maximum percent change from baseline in the PEF observed up to 2 hours following completion of dosing on study days 1 and 22. The baseline PEF was defined as the average of the test-day pre-dose baseline PEF values.
  The reason for the two primary endpoints was that FEV1 is difficult to obtain in children below 7 years of age.
Time Frame: Days 1 and 22: 30±5 and 5±2 minutes prior to dosing, and 7.5±2, 20±5, 35±5, 50±5, 65±10, 125±10 post dosing
Population: Observed cases
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
percentage change from baseline
  Day 1 (n=52, 51) | 20.040 (1.982) | 12.468 (2.004)
  Day 22 (n=51, 47) | 16.776 (1.997) | 12.994 (2.076)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1 A repeated measures mixed model, with terms for treatment, pooled center, study day, treatment by study day interaction, and baseline as a covariate, and subject as a random term, was used to make comparisons between placebo and active with respect to PEFmax%0-2 at Days 1 and 22, with observed case data; Test type: Superiority or Other; p = 0.0074, repeated measures ANOVA — significance level of 0.05; Mean Difference (Final Values) = 7.572, 95% CI 2-sided [2.077 to 13.067] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22 A repeated measures mixed model, with terms for treatment, pooled center, study day, treatment by study day interaction, and baseline as a covariate, and subject as a random term, was used to make comparisons between placebo and active with respect to PEFmax%0-2 at Days 1 and 22, with observed case data; Test type: Superiority or Other; p = 0.1843, repeated measures ANOVA — significance level of 0.05; Mean Difference (Final Values) = 3.782, 95% CI 2-sided [-1.832 to 9.397] — Active - Placebo

5. Secondary Outcome: Baseline Adjusted Area-under-the-Effect Curve for Percent of Predicted Forced Expiratory Volume in One Second (FEV1) Over 6 Hours Post-dose on Day 22 Using Both Day 1 and Day 22 Baselines
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters. Values are then expressed as the percentage of FE1 values predicted for a 'normal' population. Predicted FEV1 values were computed and adjusted for age, height and gender according to Eigen et al. for subjects 4-5 years of age and to Quanjer et al. for subjects aged 6-11 years using American Thoracic Society (ATS) criteria.
  The area under-the-effect curves for percent-predicted FEV1 were calculated according to the trapezoidal rule and were based on actual (not scheduled) measurement times.
Time Frame: Baseline (Day 1 or Day 22: 35±5 and 10±2 minutes prior to dosing), Day 22 (5±2, 15±5, 30±5, 45±5, 60±10, 120±10, 240±10, and 360±10 minutes post-dosing or last observation)
Population: Intent-To-Treat (ITT) population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: Percent of Predicted FEV1 * Hours
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
Percent of Predicted FEV1 * Hours
  Day 22 Baseline (n=52, 51) | 31.046 (3.531) | 21.338 (3.588)
  Day 1 Baseline (n=51, 51) | 25.060 (6.748) | 24.167 (6.773)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 22 Baseline; Test type: Superiority or Other; p = 0.0507, ANCOVA — significance level of 0.05; terms for treatment and center, baseline as a covariate; Mean Difference (Final Values) = 9.707, 95% CI 2-sided [-0.030 to 19.445] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 1 Baseline; Test type: Superiority or Other; p = 0.9240, ANOVA — significance level of 0.05; terms for treatment and center; Mean Difference (Final Values) = 0.892, 95% CI 2-sided [-17.634 to 19.419] — Active - Placebo

6. Secondary Outcome: Baseline-Adjusted Area-under-the Effect Curve for Peak Expiratory Flow (PEF) Over 6 Hours Post-dose on Day 22 Using Both Day 1 and Day 22 Baselines
Description: The PEF test is conducted by having a person blow as hard as they can into a mouthpiece attached to a sensor that measures the rate of air blown.
  The area under-the-effect curves for PEF were calculated according to the trapezoidal rule and were based on actual (not scheduled) measurement times.
Time Frame: Baseline (Day 1 or Day 22: 30±5 and 5±2 minutes prior to dosing Day 22: 7.5±2, 20±5, 35±5, 50±5, 65±10, 125±10 post dosing or last observation
Population: Intent-To-Treat (ITT) population with Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: Liters/Minute*Hours
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
Liters/Minute*Hours
  Day 22 Baseline (n=52, 51) | 120.82 (17.486) | 90.693 (17.753)
  Day 1 Baseline (n=52, 51) | 139.42 (25.782) | 96.842 (26.117)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 22 Baseline; Test type: Superiority or Other; p = 0.2186, ANCOVA — significance level of 0.05; terms for treatment and center, baseline as a covariate; Mean Difference (Final Values) = 30.124, 95% CI 2-sided [-18.169 to 78.417] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 1 Baseline; Test type: Superiority or Other; p = 0.2375, ANCOVA — significance level of 0.05; terms for treatment and center, baseline as a covariate; Mean Difference (Final Values) = 42.578, 95% CI 2-sided [-28.541 to 113.70] — Active - Placebo

7. Secondary Outcome: Maximum Percent-Predicted FEV1 (Max PPFEV1, %) Observed up to Two Hours Following Completion of Dosing on Study Days 1 and 22 (Observed Case)
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters. Values are then expressed as the percentage of FE1 values predicted for a 'normal' population. Predicted FEV1 values were computed and adjusted for age, height and gender according to Eigen et al. for subjects 4-5 years of age and to Quanjer et al. for subjects aged 6-11 years using American Thoracic Society (ATS) criteria.
Time Frame: Days 1 and 22: 5±2, 15±5, 30±5, 45±5, 60±10, 120 ±10 post dosing
Population: Observed cases (i.e. available data only)
Measure: Mean (Standard Error); unit: percentage of predicted FEV1
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 51 | 51
percentage of predicted FEV1
  Day 1 (n=51, 51) | 95.898 (1.451) | 89.374 (1.462)
  Day 22 (n=51, 47) | 94.650 (1.451) | 90.652 (1.488)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.0017, ANOVA — significance level of 0.05; terms for treatment, center, time, time x treatment, subject as a random; Mean Difference (Final Values) = 6.524, 95% CI 2-sided [2.524 to 10.523] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.0521, ANOVA — significance level of 0.05; terms for treatment, center, time, time x treatment, subject as a random; Mean Difference (Final Values) = 3.998, 95% CI 2-sided [-0.037 to 8.032] — Active - Placebo

8. Secondary Outcome: Time To Maximum Forced Expiratory Volume in One Second (FEV1) Over Six Hours Post-Dose On Days 1 and 22
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters.
  Time to maximum FEV1 is defined as the number of minutes required for the baseline FEV1 to increase to the highest FEV1 post dose during the 6 hour observation period.
  Median time and confidence intervals obtained via separate Kaplan-Meier estimates for each study day.
Time Frame: Days 1 and 22: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5, 45±5, 60±10, 120 ±10 post dosing
Population: Intent-To-Treat (ITT) population; Last Observation Carried Forward (LOCF) used for Day 22
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
minutes
  Day 1 (n=51, 51) | 43.95 [32.03 to 51.73] | 45.25 [30.32 to 62.82]
  Day 22 with LOCF (n=52, 51) | 41.54 [29.55 to 45.67] | 61.05 [46.53 to 120.7]
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.0647, Regression, Cox — significance level of 0.05; Cox Proportional Hazard = 1.477, 95% CI 2-sided [0.98 to 2.23] — Active/Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.0005, Regression, Cox — significance level of 0.05; Cox Proportional Hazard = 2.088, 95% CI 2-sided [1.38 to 3.15] — Active/Placebo

9. Secondary Outcome: Time To Maximum Peak Expiratory Flow (PEF) Over Six Hours Post-Dose On Days 1 and 22
Description: The PEF test is conducted by having a person blow as hard as they can into a mouthpiece attached to a sensor that measures the rate of air blown.
  Time to maximum PEF is defined as the number of minutes required for the baseline PEF to increase to the highest PEF post-dose for the 6 hour observation period. Median time and confidence intervals obtained via separate Kaplan-Meier estimates for each study day.
Time Frame: Days 1 and 22: 30±5 and 5±2 minutes prior to dosing, and 7.5±2, 20±5, 35±5, 50±5, 65±10, 125±10 post dosing
Population: ITT population; Last Observation Carried Forward (LOCF) used for Day 22
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
minutes
  Day 1 (n=52, 51) | 41.50 [34 to 64] | 35.00 [33 to 65]
  Day 22 with LOCF (n=52, 51) | 34.5 [22 to 50] | 63.00 [35 to 115]
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.5059, Regression, Cox — significance level of 0.05; Cox Proportional Hazard = 1.141, 95% CI 2-sided [0.77 to 1.69] — Active/Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.0333, Regression, Cox — significance level of 0.05; Cox Proportional Hazard = 1.533, 95% CI 2-sided [1.03 to 2.27] — Active/Placebo

10. Secondary Outcome: Participant Responses: Percentage of Participants With a >=15% Increase in Baseline FEV1 Within 30 Minutes Post-Dose on Days 1 and 22
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters. This outcome counts participants who responded to therapy by obtaining a >+15% increase in FEV1 within 30 minutes of dose.
  The baseline FEV1 was defined as the average of the two test-day pre-dose baseline FEV1 values.
Time Frame: Days 1 and 22: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5 post dosing
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 51 | 51
percentage of participants
  Day 1 (n=51, 51) | 17.6 | 9.8
  Day 22 (n=51, 47) | 17.6 | 6.4
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.3888, Fisher Exact — significance level of 0.05
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.1249, Fisher Exact — significance level of 0.05

11. Secondary Outcome: Participant Responses: Percentage of Participants With a >=12% Increase in Baseline FEV1 Within 30 Minutes Post-Dose on Days 1 and 22
Description: The FEV1 test is conducted by having a person empty their lungs of air into a mouthpiece attached to a sensor that measures the amount of air blown measured in liters. This outcome counts participants who responded to therapy by obtaining a >+12% increase in FEV1 within 30 minutes of dose.
  The baseline FEV1 was defined as the average of the two test-day pre-dose baseline FEV1 values.
Time Frame: Days 1 and 22: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5 post dosing
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 51 | 51
percentage of participants
  Day 1 (n=51, 51) | 33.3 | 13.7
  Day 22 (n=51, 47) | 29.4 | 14.9
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.0343, Fisher Exact — significance level of 0.05
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.0962, Fisher Exact — significance level of 0.05

12. Secondary Outcome: Participant Responses: Percentage of Participants With a >=15% Increase in Baseline PEF Within 30 Minutes Post-Dose on Days 1 and 22
Description: The PEF test is conducted by having a person blow as hard as they can into a mouthpiece attached to a sensor that measures the rate of air blown. This outcome counts participants who responded to therapy by obtaining a >+15% increase in PEF within 30 minutes of dose.
  The baseline PEF was defined as the average of the two test-day pre-dose baseline PEF values.
Time Frame: Days 1 and 22: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5 post dosing
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
percentage of participants
  Day 1 (n=52, 51) | 44.2 | 19.6
  Day 22 (n=51, 47) | 41.2 | 23.4
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.0109, Fisher Exact — significance level of 0.05
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.0845, Fisher Exact — significance level of 0.05

13. Secondary Outcome: Participant Responses: Percentage of Participants With a >=12% Increase in Baseline PEF Within 30 Minutes Post-Dose on Days 1 and 22
Description: The PEF test is conducted by having a person blow as hard as they can into a mouthpiece attached to a sensor that measures the rate of air blown. This outcome counts participants who responded to therapy by obtaining a >+12% increase in PEF within 30 minutes of dose.
  The baseline PEF was defined as the average of the two test-day pre-dose baseline PEF values.
Time Frame: Days 1 and 22: 35±5 and 10±2 min prior to dosing, and at 5±2, 15±5, 30±5 post dosing
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
percentage of participants
  Day 1 (n=52, 51) | 57.7 | 25.5
  Day 22 (n=51, 47) | 56.9 | 29.8
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Day 1; Test type: Superiority or Other; p = 0.0013, Fisher Exact — significance level of 0.05
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Day 22; Test type: Superiority or Other; p = 0.0085, Fisher Exact — significance level of 0.05

14. Secondary Outcome: Weekly Average Highest (Worst) Daily Asthma Symptom Scores for Weeks 1, 2 and 3
Description: Highest daily asthma symptom scores by study week. For this assessment, patients self-evaluate and record on the diary card the following asthma symptoms experienced during the day (i.e. last 12-14 hours): wheeze, shortness of breath, cough, tightness of chest. The worst of these symptoms were scored daily on a four-point scale:
  * 0 = No symptoms occurred
  * 1 = Symptom occurred but did not interfere with daily activity
  * 2 = Symptom occurred but was sometimes annoying or interfered with daily activity
  * 3 = Symptom present even at rest and was annoying or interfered with daily activity
Time Frame: Weeks 1, 2, 3
Population: ITT population.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
units on a scale
  Week 1 (N=50, N=50) | 0.370 (0.070) | 0.442 (0.070)
  Week 2 (N=50, N=49) | 0.376 (0.070) | 0.547 (0.071)
  Week 3 (N=47, N=48) | 0.336 (0.072) | 0.474 (0.071)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Week 1; Test type: Superiority or Other; p = 0.4674, ANCOVA — significance level of 0.05; terms for treatment, center, week, week by treatment, baseline as a covariate, subject as random; Mean Difference (Final Values) = -0.072, 95% CI 2-sided [-0.265 to 0.122] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Week 2; Test type: Superiority or Other; p = 0.0840, ANCOVA — significance level of 0.05; terms for treatment, center, week, week by treatment, baseline as covariate, subject as random; Mean Difference (Final Values) = -0.171, 95% CI 2-sided [-0.365 to 0.023] — Active - Placebo
Statistical Analysis 3: Comparison: Albuterol vs Placebo; Week 3; Test type: Superiority or Other; p = 0.1699, ANCOVA — significance level of 0.05; terms for treatment, center, week, week by treatment, baseline as covariate, subject as random; Mean Difference (Final Values) = -0.138, 95% CI 2-sided [-0.335 to 0.059] — Active - Placebo

15. Secondary Outcome: The Number of Asthma-Related Nocturnal Awakenings Per Week Requiring the Use of Rescue Medication
Description: Participants recorded every morning on awakening the number of asthma-related nocturnal awakenings requiring use of rescue medication that occurred during the previous night.
Time Frame: Run-in (Days -21 to -1), Weeks 1, 2, 3
Population: ITT population
Measure: Mean (Standard Deviation); unit: awakenings/week
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
awakenings/week
  Run-In (N=52, N=51) | 1.15 (2.97) | 1.06 (2.44)
  Week 1 (N=51, N=50) | 1.14 (3.25) | 1.00 (2.84)
  Week 2 (N=51, N=49) | 1.16 (3.82) | 0.73 (1.97)
  Week 3 (N=49, N=48) | 0.65 (2.21) | 1.33 (3.13)

16. Secondary Outcome: Weekly Average Peak Expiratory Flow (PEF) Obtained Pre-Dose Each Morning
Description: Participants measured their PEF as trained by taking as deep a breath as possible, placing their mouth firmly around the mouthpiece of the flow meter to form a tight seal, and exhaling as hard and as fast as possible. Subjects repeated the process twice at intervals of approximately 30 seconds, and then recorded the highest of the three PEF values on the diary card.
Time Frame: Weeks 1, 2, 3
Population: ITT population
Measure: Mean (Standard Error); unit: Liters/minute
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
Liters/minute
  Week 1 (N=51, N=50) | 229.65 (4.800) | 219.72 (4.854)
  Week 2 (N=51, N=49) | 229.90 (4.800) | 218.97 (4.870)
  Week 3 (N=49, N=48) | 231.28 (4.820) | 221.73 (4.880)
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Week 1; Test type: Superiority or Other; p = 0.1391, ANCOVA — significance level of 0.05; terms for treatment, center, week, week by treatment, baseline as a covariate, subject as random; Mean Difference (Final Values) = 9.926, 95% CI 2-sided [-3.256 to 23.108] — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Week 2; Test type: Superiority or Other; p = 0.1043, ANCOVA — significance level of 0.05; terms for treatment, center, week, week by treatment, baseline as a covariate, subject as random; Mean Difference (Final Values) = 10.923, 95% CI 2-sided [-2.278 to 24.124] — Active - Placebo
Statistical Analysis 3: Comparison: Albuterol vs Placebo; Week 3; Test type: Superiority or Other; p = 0.1570, ANCOVA — significance level of 0.05; terms for treatment, center, week, week by treatment, baseline as a covariate, subject as random; Mean Difference (Final Values) = 9.546, 95% CI 2-sided [-3.705 to 22.798] — Active - Placebo

17. Secondary Outcome: Weekly Average Number of Puffs of Rescue Medication Taken Each Day for Study Weeks 1, 2 and 3
Description: Participants recorded every morning on awakening the number of asthma-related nocturnal awakenings requiring use of rescue medication that occurred during the previous night and the number of puffs of rescue albuterol used during the night after going to bed. At the end of each day, the number of puffs of albuterol rescue medication used during the day were recorded.
Time Frame: Weeks 1, 2, 3
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: Number of puffs per day
Arm/Group | Albuterol | Placebo
Number analyzed (Participants) | 52 | 51
Number of puffs per day
  Week 1 (N=51, N=50) | 0.074 [0.009 to 0.138] | 0.075 [0.011 to 0.139]
  Week 2 (N=51, N=49) | 0.084 [0.011 to 0.158] | 0.088 [0.013 to 0.163]
  Week 3 (N=49, N=48) | 0.078 [0.010 to 0.146] | 0.088 [0.013 to 0.163]
Statistical Analysis 1: Comparison: Albuterol vs Placebo; Week 1 P-value, mean and confidence interval calculated from a 0 inflated mixed poisson regression model with fixed effect terms for treatment, week, treatment by week interaction, baseline as a covariate and a random term for subject. The null hypothesis is that the ratio equals 1. Estimated means are conditional upon the random effect, assume a random effect of 0 and a covariate value at the average; Test type: Superiority or Other; p = 0.9846, mixed poisson regression model — significance level of 0.05; ratio of Active to Placebo = 0.989, 95% CI 2-sided [-0.121 to 2.099]
Statistical Analysis 2: Comparison: Albuterol vs Placebo; Week 2 P-value, mean and confidence interval calculated from a 0 inflated mixed poisson regression model with fixed effect terms for treatment, week, treatment by week interaction, baseline as a covariate and a random term for subject. The null hypothesis is that the ratio equals 1. Estimated means are conditional upon the random effect, assume a random effect of 0 and a covariate value at the average; Test type: Superiority or Other; p = 0.9447, mixed poisson regression model — significance level of 0.05; ratio of Active to Placebo = 0.961, 95% CI 2-sided [-0.116 to 2.039]
Statistical Analysis 3: Comparison: Albuterol vs Placebo; Week 3 P-value, mean and confidence interval calculated from a 0 inflated mixed poisson regression model with fixed effect terms for treatment, week, treatment by week interaction, baseline as a covariate and a random term for subject. The null hypothesis is that the ratio equals 1. Estimated means are conditional upon the random effect, assume a random effect of 0 and a covariate value at the average; Test type: Superiority or Other; p = 0.8326, mixed poisson regression model — significance level of 0.05; ratio of Active to Placebo = 0.887, 95% CI 2-sided [-0.111 to 1.885]

ADVERSE EVENTS:
Time Frame: Days 1-22
Groups:
- Albuterol: Albuterol-HFA-MDI 180 mcg, four times a day
Arm/Group | Albuterol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 7/52 | 5/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol (N=52) | Placebo (N=51)
Nasopharyngitis (Infections and infestations) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If review shows that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for up to 90 additional days to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure of multicenter data, but not longer than 12 months from study completion/termination at all participating sites.